CLINICAL TRIAL: NCT03741296
Title: REVISITS Trial: Revision Single or Two Stage Surgery for Periprosthetic Hip Infection - a Multicentre Randomized Clinical Trial
Brief Title: REVISITS: Revision Single or Two Stage Surgery
Acronym: REVISITS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-0278
Record Dates: First submitted 2018-11-07; First posted 2018-11-14 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Total Hip Replacement; Arthroplasty Complications
Keywords: Hip replacement; periprosthetic hip infection; single stage revision; two-stage revision

STUDY DESIGN:
Intervention Model Description: This is a study is a multicentre, prospective, parallel, two-arm, randomized controlled trial aiming to assess the efficacy of single stage revision peri-prosthetic joint infection of hip arthroplasty in adult's patients, compared to the current gold standard of care, two-stage revision.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- single stage revision (Active Comparator): One surgery where the infected artificial joint will be removed along with all components, cement, and any potentially infected material. The surgical site will be debrided and washed out before a new artificial hip joint (prosthesis) is implanted. All the procedures will be done in a single surgery.
  Interventions: Procedure: Single stage revision
- two-stage revision (Active Comparator): Patients will undergo 2 separated surgeries. In the first operation, the infected artificial joint will be removed along with all components, cement, and any potentially infected material. The surgical site will be debrided, washed out and a spacer will be placed in the hip (temporarily replace prosthesis).
  A secondary surgery to re-implant the hip will be performed with an interval period of 4-10 weeks when the infection is cleared.
  The site will be debrided and irrigated, and any component/spacer will be removed. A new artificial joint will then be implanted.
  Interventions: Procedure: Two-stage revision

INTERVENTIONS:
Procedure: Single stage revision — One-stage exchange hip joint replacement surgery
  Arms: single stage revision
Procedure: Two-stage revision — Two-stage exchange hip joint replacement surgery
  Arms: two-stage revision

SUMMARY:
Hip replacement surgery is common, with over 60,000 cases in Canada annually. After hip replacement, about 1-2% patients develop a deep infection in their artificial hip implant, called a periprosthetic joint infection (PJI). It can results in severe pain, disability and death.

There are two types of surgical treatment: a single-stage revision that involves removing the joint, thoroughly cleaning the infected area and implanting a new joint, all in the same surgical procedure; a two-stage revision involves removing the joint, waiting at least 8 weeks while treating the patients with antibiotics and then doing re-implantation of the joint.

DETAILED DESCRIPTION:
Peri-prosthetic infection is an uncommon but severe complication of joint replacement (arthroplasty) with a reported rate between 0.6 to 2.2%. Although the likelihood of infection is relatively small, the psychological and economic impact, as well as long-term implications to both the patient and healthcare system, can be catastrophic.

The current gold standard treatment for peri-prosthetic infection is a two-stage strategy, where the artificial hip joint is removed and a new replacement delayed for at least 8 weeks until clear evidence of infection eradication is obtained. During this time the patient may be non-ambulatory, non- or partial-weight bearing and then a wait for re-listing for the second surgery.

An alternative treatment that has recently been more widely used is to perform a single stage revision. That involves removing the implants and then irrigating and debriding and finally implanting the new replacements prostheses. This is all done in one surgery. The advantage of this technique is that there is only one procedure and usually the patient is allowed to bear weight on the joint.

Primary Objective:

To compare pain and physical function assessed by the Oxford hip score, between the single and two-stage revision surgery for a periprosthetic hip infection in adults

Secondary Objectives:

To compare pain, function, quality of life, rates of reinfection, complications, cost-effectiveness and health economic impact.

Tertiary Objectives:

To involve building partnerships between patients, researchers and clinicians. Patients will be engaged in the trial development and knowledge translation.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged 18 years or above
* A clinical diagnosis of deep hip periprosthetic joint infection according to the Musculoskeletal Infection Society criteria
* Require revision surgery (either single-or two-stage revision) for hip periprosthetic joint infection in the opinion of the treating consultant orthopaedic surgeon
* The patient is not a candidate for Debridement, Antibiotics and Implant Retention (DAIR) treatment with retention of the implant
* Willing and able to sign the written consent, follow the protocol and attend follow-up
* Able to read and understand English

Exclusion Criteria:

* Culture-negative infection (organism not identified)
* Patients with systemic sepsis who require emergent surgery
* Resistant organisms not sensitive to available intravenous antibiotics
* Revision surgery or previous two-stage reimplant
* Unable or unwilling to undergo either single-or two-stage revision surgery
* Cognitive impairment (dementia, Alzheimer, etc.) which will prevent patients from completing the primary outcome measure
* Medical contra-indication to surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2019-04 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Patient-reported hip function | Questionnaire will be completed by patients at 9 months after surgery
  Measured by means of the Oxford Hip Score - A short questionnaire consists of 12 questions ranging from 0 to 48 points, designed to assess function and pain after hip replacement surgery. Higher values represent a better outcome. Scores between 40-48 indicate satisfactory joint function

SECONDARY OUTCOMES:
Health status and quality of life | Questionnaire will be completed by patients before the surgery and at 6, 9, 12 and 24 months after surgery
  EuroQol-5D (EQ-5D-5L) is a questionnaire where patients self-rate their level of severity of health status and health-related quality of life. Consists of 5 dimensions (mobility, self care, usual activities, pain/discomfort, anxiety/depression) and each one of them has 5 levels (no problems, slight problems, moderate problems, severe problems, and extreme problems) where patients will indicate how they feel regarding their health status and quality of life.
Reinfection rates | will be assessed at 6 weeks, 3, 6, 9,12 and 24 months after surgery
  Recurrence of infection by the same organism or reinfection with a new organism as determined by the criteria using the Musculoskeletal Infection Society criteria.
  1. There is a sinus tract communicating with the prosthesis; or
  2. A pathogen is isolated by culture from at least two separate tissue or fluid samples obtained from the affected prosthetic joint; or
  3. Four of the following six criteria exist:
     1. Elevated serum erythrocyte sedimentation rate (ESR) and serum C-reactive protein (CRP) concentration
     2. Elevated synovial leukocyte count,
     3. Elevated synovial neutrophil percentage (PMN%)
     4. Presence of purulence in the affected joint
     5. Isolation of a microorganism in one culture of periprosthetic tissue or fluid
     6. Greater than five neutrophils per high-power field in five high-power fields observed from histologic analysis of periprosthetic tissue at 400x magnification
Patient-reported hip function | Questionnaire will be completed by patients at 12 and 24 months after surgery
  Measured by means of the Oxford Hip Score - A short questionnaire consists of 12 questions ranging from 0 to 48 points, designed to assess function and pain after hip replacement surgery. Higher values represent a better outcome. Scores between 40-48 indicate satisfactory joint function
Visual Analog Pain Scale | Pain scale will be assessed before the surgery and at 24 and 48 hours, 6 weeks, 3,6, 9, 12 and 24 months after surgery
  Assess pain from a visual scale that ranges from 0 to 10. Straight line with the endpoints defining extreme limits such as 'no pain at all' (zero) and 'pain as bad as it could be' (ten)
Hospital readmission | Will be assessed within 30 days of discharge
  If patients who were discharged after surgery have an unplanned readmission for any cause to an hospital, the reason for readmission being related or not to the surgery
Hospital length of stay | Will be assessed from admission to discharge (up to 30 days)
  The duration of a single episode of hospitalization (in days)

CONTACTS AND LOCATIONS:
Overall Officials: Amit Atrey, MD, Principal Investigator — Unity Health Toronto

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kunutsor SK, Whitehouse MR, Blom AW, Beswick AD; INFORM Team. Re-Infection Outcomes following One- and Two-Stage Surgical Revision of Infected Hip Prosthesis: A Systematic Review and Meta-Analysis. PLoS One. 2015 Sep 25;10(9):e0139166. doi: 10.1371/journal.pone.0139166. eCollection 2015. PMID 26407003
- [Background] Lopez D, Leach I, Moore E, Norrish AR. Management of the Infected Total Hip Arthroplasty. Indian J Orthop. 2017 Jul-Aug;51(4):397-404. doi: 10.4103/ortho.IJOrtho_307_16. PMID 28790468
- [Background] Kapadia BH, Berg RA, Daley JA, Fritz J, Bhave A, Mont MA. Periprosthetic joint infection. Lancet. 2016 Jan 23;387(10016):386-394. doi: 10.1016/S0140-6736(14)61798-0. Epub 2015 Jun 28. PMID 26135702
- [Background] Dale H, Fenstad AM, Hallan G, Havelin LI, Furnes O, Overgaard S, Pedersen AB, Karrholm J, Garellick G, Pulkkinen P, Eskelinen A, Makela K, Engesaeter LB. Increasing risk of prosthetic joint infection after total hip arthroplasty. Acta Orthop. 2012 Oct;83(5):449-58. doi: 10.3109/17453674.2012.733918. PMID 23083433
- [Background] Blom AW, Taylor AH, Pattison G, Whitehouse S, Bannister GC. Infection after total hip arthroplasty. The Avon experience. J Bone Joint Surg Br. 2003 Sep;85(7):956-9. doi: 10.1302/0301-620x.85b7.14095. PMID 14516026
- [Background] Phillips JE, Crane TP, Noy M, Elliott TS, Grimer RJ. The incidence of deep prosthetic infections in a specialist orthopaedic hospital: a 15-year prospective survey. J Bone Joint Surg Br. 2006 Jul;88(7):943-8. doi: 10.1302/0301-620X.88B7.17150. PMID 16799001
- [Background] Lenguerrand E, Whitehouse MR, Beswick AD, Jones SA, Porter ML, Blom AW. Revision for prosthetic joint infection following hip arthroplasty: Evidence from the National Joint Registry. Bone Joint Res. 2017 Jun;6(6):391-398. doi: 10.1302/2046-3758.66.BJR-2017-0003.R1. PMID 28642256
- [Background] Chen SY, Hu CC, Chen CC, Chang YH, Hsieh PH. Two-Stage Revision Arthroplasty for Periprosthetic Hip Infection: Mean Follow-Up of Ten Years. Biomed Res Int. 2015;2015:345475. doi: 10.1155/2015/345475. Epub 2015 Apr 29. PMID 26064901
- [Background] Kunutsor SK, Whitehouse MR, Blom AW, Board T, Kay P, Wroblewski BM, Zeller V, Chen SY, Hsieh PH, Masri BA, Herman A, Jenny JY, Schwarzkopf R, Whittaker JP, Burston B, Huang R, Restrepo C, Parvizi J, Rudelli S, Honda E, Uip DE, Bori G, Munoz-Mahamud E, Darley E, Ribera A, Canas E, Cabo J, Cordero-Ampuero J, Redo MLS, Strange S, Lenguerrand E, Gooberman-Hill R, Webb J, MacGowan A, Dieppe P, Wilson M, Beswick AD; Global Infection Orthopaedic Management Collaboration. One- and two-stage surgical revision of peri-prosthetic joint infection of the hip: a pooled individual participant data analysis of 44 cohort studies. Eur J Epidemiol. 2018 Oct;33(10):933-946. doi: 10.1007/s10654-018-0377-9. Epub 2018 Apr 5. PMID 29623671
- [Background] Kunutsor SK, Whitehouse MR, Lenguerrand E, Blom AW, Beswick AD; INFORM Team. Re-Infection Outcomes Following One- And Two-Stage Surgical Revision of Infected Knee Prosthesis: A Systematic Review and Meta-Analysis. PLoS One. 2016 Mar 11;11(3):e0151537. doi: 10.1371/journal.pone.0151537. eCollection 2016. PMID 26967645